CLINICAL TRIAL: NCT06923618
Title: Identification of Aging Biomarkers for Better Tailoring of Cancer Treatment in Older Patients With Lung Cancer: a Multicenter Clinico-biological Cohort Study
Brief Title: Cancer of the Lung And SeneScencE - Prospective Cohort 1
Acronym: CLASSE-P1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ARC Foundation and Inserm (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP241246; ID-RCB Number (Other: 2024-A02393-44)
Record Dates: First submitted 2025-02-17; First posted 2025-04-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Aging biomarkers
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood samples — Blood samples (5 ml) during surgery or within 3 days before.

SUMMARY:
The main objective is to identify and assess the predictive value of ageing and senescence biomarkers (methylome, telomeres, inflammageing) and senescent cells in tissues to improve prognosis assessment older patients with locally or locally-advanced Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Geriatric assessment allows oncologists to stratify older cancer patients into risk categories (fit, vulnerable and frail) but few patients benefit from it. Yet, they do not evaluate physiological reserves when oncologists are in dire need of quantitative tools accounting for age-related changes. This decade has witnessed the remarkable power of multiple tools (epigenetics, telomere integrity, cellular and immunosenescence) to estimate an individual's age. These tools hold the potential for routine implementation in the clinic and to be combined with existing tests. The main objective is to identify and assess the predictive value of ageing and senescence biomarkers (methylome, telomeres, inflammageing) and senescent cells in tissues to improve to improve prognosis assessment in older patients with locally or locally-advanced Non-Small Cell Lung Cancer (NSCLC).

The ambition of this study is to refine the prognosis assessment and optimize decision-making process, better anticipate adverse-events and unplanned hospitalization and better manage and care high risk patients of early death, unplanned hospitalization, major complication or toxicities and altered quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients 70 years and over
* Local or locally advanced (Clinic stage I-IIIA) NSCLC (clinically (or radiologically) suspected or histologically proven)
* Surgical Curative Intent
* Signed informed Consent (or signed by the curator or tutorship)
* Affiliated to social security administrative care service

Exclusion Criteria:

* Synchronous cancer (histologically proven or strongly suspected non-lung cancer in the 6 months prior to inclusion (excluding basal cell cancer and prostate cancer with local treatment (radiotherapy or surgery) or active surveillance without systemic treatment (chemotherapy, hormone therapy)).
* Subject deprived of liberty by judicial or administrative decision or patient under guardianship
* Subject unable to understand the purpose and conditions of the study and unable to give consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Unplanned hospitalizations within 12 months | 12 months post surgery
  Number of unplanned hospitalizations within 12 months

SECONDARY OUTCOMES:
Mortality (all-cause) and cause-specific | Month 12 and Month 60 post surgery
  Number of death (all-cause) and cause-specific at Month12 and Month 60
Surgical Complications | Month 3 and Month 6 post surgery
  Scores on the Clavien-Dindo Scale at Month 3 and Month 6
Major Toxicities | Month 3 and Month 6 post surgery
  Scores on the NCI-PRO-CTCA (National Cancer Institute Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) scale (Lickert scale with 5 levels/item) at Month 3 . A higher score means worse outcome.
Quality of Life Core 30 | Month 6 and Month 12 post surgery.
  Scores on the Quality of Life (QLQ) patients self-questionnaires Core 30 (0-100 points) at Month 6 and Month 12. A higher score means worse outcome.
Quality of Life Lung Cancer 13 | Month 6 and Month 12 post surgery
  Scores on the Quality of Life (QLQ) patients self-questionnaires Lung Cancer 13 (0-100 points) at Month 6 and Month 12. A higher score means worse outcome.
Quality of Life Elderly 14 | Month 6 and Month 12 post surgery
  Scores on the Quality of Life (QLQ) patients self-questionnaires Elderly 14 (0-100 points) at Month 6 and Month 12. A higher score means worse outcome.
Disease-free survival | Month 3, Month 12 and Month 60 post surgery
  Disease-free survival on imaging (CT scan) at Month 3, Month 6, Month 12 and Month 60
Geriatric Parameters G-CODE | Month 3 and Month 6 post surgery
  Score on Geriatric-COre Data sEt (G-CODE) (0-17) at Month 3 and Month 6. A higher score means better outcome.
Geriatric Parameters Hand grip | Month 3 and Month 6 post surgery
  Scores on Hand grip (kg) at Month 3 and Month 6. A higher score means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Florence CANOUÏ-POITRINE, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No